CLINICAL TRIAL: NCT04689308
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation and Dose Expansion Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Antitumor Activity of MH048 in Subjects With Selected Relapsed/Refractory B-cell Malignancies
Brief Title: This is a Phase 1 Study of MH048 in Patients With Selected Relapsed/Refractory B-cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minghui Pharmaceutical (Shanghai) LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MH048-CP001CN
Record Dates: First submitted 2020-12-14; First posted 2020-12-30 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Relapsed/Refractory B-cell Malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: Dose Escalation and Determination of RP2D (Experimental): Part A: Dose Escalation and determination of RP2D, multiple dose levels of MH048 to be evaluated
  Interventions: Drug: MH048
- Part B: Dose Expansion in Selected Relapsed/Refractory B-cell Malignancies (Experimental): Part B: Selected relapsed/refractory B-NHL subjects with at least 1 prior systemic OR standard-of-care therapy.
  Interventions: Drug: MH048

INTERVENTIONS:
Drug: MH048 — Soft gel capsules 5 mg and 25 mg，oral MH048 should be administered after an overnight fast.
  Other Names: MH048 Soft Gel Capsules

SUMMARY:
This is a Phase 1 study of MH048 in patients with selected Relapsed/Refractory B-cell Malignancies.

DETAILED DESCRIPTION:
This is an open-label, multi-center Phase 1 study of MH048 in patients with selected Relapsed/Refractory B-cell Malignancies.

This study includes 2 parts: Part A is the dose escalation part of the study, and Part B is the dose expansion part of the study. In Part A, patients were enrolled using accelerated titration design for the first three single patient cohorts and 3+3 dose escalation design for the rest cohorts. The starting dose of MH048 in soft gel capsule form was 5 mg/day QD. Cycle length will be 28 days. In Part B, the dose and lymphoma subtypes for expansion phase will depend on the results from Part A.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age;
2. Willing and able to understand and sign an informed consent form and to comply with all aspects of the protocol;
3. Life expectancy of ≥12 weeks;
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
5. Histologically confirmed B-cell Malignancies who have relapsed or are refractory to standard of care therapies, and have received ≥1 prior lines of therapy:

   Part A: Subjects with B-cell Malignancies (regardless of subtype); Part B: Subjects With Selected Relapsed/Refractory B-cell Malignancies based on data from Part A;
6. There must be radiographically measurable disease for effects assess at dose expansion cohort;
7. Adequate organ function, as specified below:

   Hematologic: Platelet count >65 × 10^9/L (may be posttransfusion, must one week before the first dose of starting study treatment); Hemoglobin (Hgb) ≥ 80 g/L; international normalized ratio (INR) or plasma prothrombin time (PT) ≤1.5 × ULN; absolute neutrophil count >1.0 × 10^9/L (growth factor use is allowed to bring pre-treatment neutrophils to >1.0 × 10^9 cells/L if bone marrow infiltration is involved, provided this is not within 7 days of starting study treatment); Hepatic: Total bilirubin <1.5 × upper limit normal (ULN), Total bilirubin <3 × ULN for Gilbert Syndrome; Aspartate aminotransferase (AST) and Alanine transaminase (ALT) ≤2.5 × ULN; Renal: Creatinine clearance ≥60 mL/min (as estimated by the Cockcroft-Gault equation );
8. Willing to have bone marrow biopsy/aspirate for baseline disease assessment and assessment of response to treatment;
9. Willingness of men and women of reproductive potential to observe conventional and highly effective birth control from the beginning of the study screening until 6 months after receiving the last treatment of investigational product. A fertile woman must be confirmed by a positive serum beta-human chorionic gonadotropin [β-hCG] test before 7 days of starting study treatment.

Exclusion Criteria:

1. History of other active malignancies within 1 years of study entry, with the exception of adequately treated in-situ carcinoma of cervix, localized basal cell or squamous cell carcinoma of skin, previous malignancy that was not recurred in 5 years;
2. History of allogeneic or autologous stem cell transplant or chimeric antigen receptor-modified T-cell (CAR-T) therapy within the past 100 days before starting study treatment, or diagnosis of graft vs host disease;
3. Clinically significant, uncontrolled cardiac or cardiovascular disease, or history of myocardial infarction, New York Heart Association (NYHA) Class III or IV, QTc prolongation (defined as a QTc > 450 ms) or other significant electrocardiogram (ECG) abnormalities including 2nd degree atrioventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min) ,within 6 months prior to planned start of MH048 treatment;
4. Transformation (e.g., Richter's transformation, prolymphocytic leukemia, or blastoid lymphoma) prior to the planned start of MH048 treatment;
5. Subjects with known or suspected history of allergy to MH048 capsules or excipients;
6. Any unresolved toxicities from prior therapy of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v5.0) Grade 2 or higher at the time of starting MH048 treatment, with the exception of toxicities not considered a safety risk (eg, alopecia, neuropathy, or asymptomatic laboratory abnormalities);
7. Active uncontrolled systemic bacterial, viral, fungal, or parasitic infection;
8. Active uncontrolled autoimmune disease;
9. Clinically significant active malabsorption syndrome;
10. Subjects with human immunodeficiency virus (HIV) , Active hepatitis B virus (HBsAg positive, or HBsAg negative/HBcAb positive ，and HBV DNA>10^3) or Active HCV infection (HCVAb positive ,and HCV RNA positive);
11. Major surgery within 4 weeks prior to planned start of MH048 treatment (expect for biopsy, laser eye surgery)；
12. Women of childbearing potential who are pregnant or lactating;
13. Subjects requiring therapeutic anticoagulation;
14. Radiotherapy with a limited field of radiation for palliation within 7 days of the first dose of MH048 treatment;
15. Received a CYP3A4, CYP2A8 strong inhibitor or inducer within 5 half-lives of planned investigational product administration；
16. Medical history of massive bleeding (hemophilia or other disease need the treatment of blood transfusion）;
17. Severe neurological/mental illness, and in the opinion of the Investigator, is unable to adhere to the requirements of the study;
18. Receipt of any investigational agent or clinical study within 28 days;
19. Unstable brain metastasis patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence and severity of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to approximately 24 Months
  Assess incidence and severity of treatment-emergent adverse events as determined by CTCAE v5.0
To determine the MTD of MH048 | At the end of Cycle 1( 28 day) of each dose escalation cohort.
  If 2 or more treated subjects at a dose level experience a DLT before Day 28, dose escalation will stop and the prior dose level will be considered the MTD for that schedule.
To establish the RP2D. | Up to approximately 24 Months
  The determination of RP2D for phase 2 according to the result of dose expansion cohorts.

SECONDARY OUTCOMES:
Characterization of Pharmacokinetics (Cmax) | At the end of Cycle 1 (each cycle is 28 days)
  Maximum drug concentration (Cmax)
Characterization of Pharmacokinetics (AUC) | At the end of Cycle 1 (each cycle is 28 days)
  Area Under the Curve (AUC)
Characterization of Pharmacokinetics (CL) | At the end of Cycle 1 (each cycle is 28 days)
  Clearance (CL)
Characterization of Pharmacokinetics (t1/2) | At the end of Cycle 1 (each cycle is 28 days)
  Elimination half-life (t1/2)
Preliminary evidence of anti-tumor activity, in terms of Objective Response Rate (ORR) | From date of enrollment until the date of best overall response (BoR) of CR or PR, assessed up to approximately 24 months.
  The number (%) of subjects with best overall response (BoR) of CR or PR.
Preliminary evidence of anti-tumor activity, in terms of Duration of Response (DOR) | From the first documented of CR or PR to the first documented PD or death due to any cause, whichever came first, , assessed up to approximately 24 months.
  The duration from the first documentation of CR or PR to the first documented PD or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, MD, Principal Investigator — 79 Qingchun Road, Shangcheng District, Hangzhou, Zhejiang, China
Locations (1):
- the First Affiliated Hospita，Medicine School of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No